CLINICAL TRIAL: NCT03977753
Title: Study to Evaluate the Efficacy of 2LVERU® JUNIOR and 2LVERU® on the Treatment of Warts.
Brief Title: Randomized, Placebo-controlled, Double Blind Study to Evaluate the Efficacy of 2LVERU®JUNIOR and 2LVERU® on the Treatment of Warts
Acronym: EVAsION
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Labo'Life (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LLB-2019-02
Record Dates: First submitted 2019-06-04; First posted 2019-06-06 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Common Wart; Flat Wart; Plantar Wart
MeSH Terms: conditions — Warts

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double-blind study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2LVERU®/2LVERU® JUNIOR (Experimental): Group N°1: 2LVERU® or 2LVERU® JUNIOR treatment (6 months of treatment)
  Interventions: Drug: 2LVERU® or 2LVERU® JUNIOR
- Placebo (Placebo Comparator): Group N°2: Placebo treatment (6 months of treatment)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 2LVERU® or 2LVERU® JUNIOR — The treatment schema consists in taking the content of one capsule a day, 15-30 minutes before breakfast, on an empty stomach, sequentially, according to capsules' numerical order: 1 through 10. When capsule number 10 is taken, capsule 1 of the next blister should be taken on the next day to continue the treatment.
  The duration of treatment will be 6 months of continuous intake of the content of 1 capsule/day.
  Arms: 2LVERU®/2LVERU® JUNIOR
Drug: Placebo — The treatment schema consists in taking the content of one capsule a day, 15-30 minutes before breakfast, on an empty stomach, sequentially, according to capsules' numerical order: 1 through 10. When capsule number 10 is taken, capsule 1 of the next blister should be taken on the next day to continue the treatment.
  The duration of treatment will be 6 months of continuous intake of the content of 1 capsule/day.
  Arms: Placebo

SUMMARY:
Human papillomavirus (HPV) infection is very common, as most people will experience infection during their lifetime. The most common manifestation of HPV infection is common warts. Common warts may appear at any age.

Conventional treatments can be used to treat warts and they are based on two mechanisms: stimulation of cellular immunity against HPVs or destruction of the lesion. These treatments are based on the location of the wart and the degree of the symptoms.

No specific antiviral therapy is available to cure warts and today, there is no treatment that allows the definitive eradication of the virus.

The 2LVERU® has been available for more than 20 years, and has received a marketing authorization in Belgium by the Federal Agency for Medicines and Health Products (FAMHP). It is used as an immune regulator in the treatment of common warts (verruca vulgaris), flat warts (verruca plana) or plantar warts (verruca plantaris) caused by Human Papillomavirus. Since 2LVERU® has been made available, clinical observational data collected on treated patients have shown the beneficial effect on the disappearance of warts.

The purpose of this placebo-controlled, randomized, double-blind trial is the comparison of the efficacy of the treatment on the disappearance of warts at the end of treatment (6-month visit) between the 2LVERU® JUNIOR and 2LVERU® versus the placebo group.

DETAILED DESCRIPTION:
The study duration will be maximum 45 months with 36 months of inclusion and 9 months of follow-up.

Patients aged 3 years and older who present common warts (Verruca vulgaris), and/or plantar warts (Verruca plantaris), and/or flat warts (Verruca plana) during a visit with their dermatologist/general practitioner.

The total number of patients to include will be 162.

Primary objective:

Comparison of the efficacy of the treatment on the disappearance of warts at the end of treatment (6-month visit) between the 2LVERU® JUNIOR and 2LVERU® versus the placebo group.

Secondary objectives

* Comparison of the efficacy of the treatment on the disappearance of warts at 4 months between groups.
* Comparison of the efficacy of the treatment on the level of disappearance (4 levels) of warts at 4 months and 6 months (end of the treatment) between groups
* Comparison of the efficacy of the treatment on the recurrence of warts 3 months after the end of treatment between groups
* Compare the pain related to warts during the study between groups
* Safety issues.

Treatment phase:

* Group n°1 = 2LVERU® JUNIOR / 2LVERU® (6 months of treatment)
* Group n°2 = Placebo (6 months of treatment)

Post-treatment Follow-up phase: 3 months

Treatment will be considered successful if the following three criteria are met for all treated warts as described at the baseline visit:

* Normal skin colour at the wart site
* Normal skin texture at the wart site
* Normal touch at the wart site Treatment will be considered a failure, at the end of the treatment, if at least one of the above three criteria is not met for all treated warts as described at the baseline visit.

ELIGIBILITY:
Inclusion Criteria:

* Patients, male or female, aged 3 years and older,
* Patients with common warts (Verruca vulgaris), and/or plantar warts (Verruca plantaris), and/or flat warts (Verruca plana),
* Patients (and/or parents if necessary) having the faculties to understand and respect the constraints of the study,
* Signature of the Informed Consent Form by the patient (and/or parents if necessary).

Exclusion Criteria:

* Patients who have received any curative warts treatment in the previous 2 months prior to the study,
* Patients who have received any homeopathic treatment in the previous 2 months prior to the study,
* Patients under immunosuppressive treatment,
* Patients having received immunotherapy or micro-immunotherapy during the last 6 months,
* Patients with known lactose intolerance,
* Pregnant or breastfeeding women,
* Patients who participated in a clinical study in the previous 2-months period,
* Patients (and/or parents of patients if necessary) who are not sufficiently motivated to engage on the total study follow-up period, or likely to travel or to move before the end of the study,
* Patients with severe immunodeficiency disease requiring long term treatment (*) or patients under chemotherapy or radiotherapy,
* Patients under listed homeopathic or phytotherapy treatment (see protocol),
* Patients addicted to or using recreational drugs,
* Patient under guardianship and/or curators, (*) important renal or respiratory insufficiency, transplanted or grafted patients, HIV/AIDS, terminal cancer.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2020-02-17 (Actual); Primary Completion 2026-12-16 (Estimated); Study Completion 2027-03-16 (Estimated)

PRIMARY OUTCOMES:
Disappearance of warts at the end of treatment (6-month visit) | 6 months
  A wart will be considered as disappeared if the colour and texture of the skin has returned to normal and can no longer be felt to the touch.

SECONDARY OUTCOMES:
Disappearance of warts at 4 months. | 4 months
Disappearance level (total disappearance, partial disappearance (50%), no modification, increase of number of warts) at 4 months | 4 months
Warts recurrence at 9 months | 9 months
Pain evaluation during the study by visual analogic scale and consumption of antalgic medication. | 6 months
  Minimum value: 0 (better outcome) Maximum Value: 10 (worse outcome)
Safety: occurence of adverse events (AEs) and severe adverse events (SAEs), considered as related or not to the study drug. | 6 months
Disappearance level (total disappearance, partial disappearance (50%), no modification, increase of number of warts) at 6 months | 6 months

CONTACTS AND LOCATIONS:
Locations (17):
- Belgium (17):
  - Private Practice, Arlon
  - Clinique Saint-Luc (Bouge), Bouge
  - Private Practice, Brussels
  - Private Practice, Écaussinnes-d'Enghien
  - Private Practice, Fontaine l'Êveque
  - Private Practice, Ghent
  - Private Practice, Gozée
  - Private Practice, Hamme-Mille
  - Private Practice, Juprelle
  - Private Practice, Mons
  - Private Practice, Namur
  - Private Practice, Oisquercq
  - Private Practice, Plancenoit
  - Private Practice, Quiévrain
  - Private Practice, Saint-Symphorien
  - Private Practice, Seneffe
  - Private Practice, Wavre

IPD SHARING:
Plan to Share IPD: No